CLINICAL TRIAL: NCT01931982
Title: Effect of GLP-1 on Microvascular Myocardial Function in Patients With Type 2
Brief Title: Effect of Glucagon-like Peptide 1 (GLP-1) on Microvascular Myocardial Function in Patients With Type 2 Diabetes.
Acronym: EGOFIP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Mette Zander, MD, PhD, Bispebjerg Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: eudraCT: 2012-005013-38; 2012-005013-38 (EudraCT Number)
Record Dates: First submitted 2013-08-20; First posted 2013-08-30 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Type 2 Diabetes; Microvascular Dysfunction
Keywords: diabetes, GLP-1, Victoza, CFR, microvascular dysfunction
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- victoza (Active Comparator): The study is a cross over study. Patients randomised to start with victoza are treated with victoza for 10 weeks. After a wash out period of 2 weeks they cross over to 10 weeks of no treatment
  Interventions: Drug: Victoza
- No treatment (No Intervention)

INTERVENTIONS:
Drug: Victoza
  Arms: victoza

SUMMARY:
The purpose of the study is to determine if a GLP-1 agonist improves microvascular perfusion in the heart of patients with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes on monotherapy with metformin or sulfonylurea or combination therapy of metformin and sulfonylurea.
* Age: 25-75 years
* BMI>25 kg/m2
* HbA1c 6,0-10 %

Exclusion Criteria:

* Current treatment with insulin or Dipeptidyl peptidase IV inhibitor.
* Haemoglobin < 6.5 mmol/l
* Documented significant stenosis of the left anterior descending artery (LAD) at coronary angiography or CT-angiography or regional dysfunction documented during dipyridamol stress-echocardiography. If stress test at baseline shows significant stenosis the patient will be excluded from the study.
* Allergy towards victoza ® (liraglutide ), Dipyridamol, Nitroglycerin or rescue medicine: Theophyllin
* Pregnancy
* Severe asthma
* Active cancer
* Severe co-morbidity with limited life-expectancy
* Estimated glomerular filtration rate (eGFR) <60 (measured at baseline)
* Severe hepatic co-morbidity
* Chronic alcohol abuse
* Heart failure with a left ventricular ejection fraction </= 45%
* Atrial fibrillation
* Chronic or previous acute pancreatitis
* Inflammatory bowel disease.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in coronary flow reserve (CFR) | CFR is measured at baseline and after 10 weeks of intervention
  CFR can be reliably assessed non-invasively by trans-thoracic Doppler flow echocardiography of the left anterior descending artery with a success rate of over 90% even in an obese population with a relative poor acoustic window. CFR is the ratio of flow during stress to during rest.

SECONDARY OUTCOMES:
Change in Endothelial function: | Endothelial function is measured at baseline and after 10 weeks of intervention
  Measurement of Peripheral Arterial Tone, with the use of the commercially available machine (Endo-PAT2000®) assesses the control of digital vascular tone by the sympathetic nervous system and nitric oxide (NO).

OTHER OUTCOMES:
Changes in HbA1c | Measurements at baseline and after 10 weeks of intervention
Change in fasting C-peptide | C-peptide is measured at baseline and after 10 weeks of intervention
Change in fasting insulin | Fasting insulin is measured at baseline and after 10 weeks of intervention
Change in fasting glucose | Fasting glucose is measured at baseline and after 10 weeks of intervention
Change in weight | Weight is measured at baseline and after 10 weeks of intervention
Change in waist circumference | Waist circumference is measured at baseline and after 10 weeks of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mette Zander, consultant, Principal Investigator — Department of Endocrinology, Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Capital Region, Denmark

REFERENCES:
- [Derived] Faber R, Zander M, Pena A, Michelsen MM, Mygind ND, Prescott E. Effect of the glucagon-like peptide-1 analogue liraglutide on coronary microvascular function in patients with type 2 diabetes - a randomized, single-blinded, cross-over pilot study. Cardiovasc Diabetol. 2015 Apr 22;14:41. doi: 10.1186/s12933-015-0206-3. PMID 25896352